CLINICAL TRIAL: NCT00132340
Title: Deep Brain Stimulation of the Globus Pallidus Interna or the Subthalamic Nucleus for Treatment of Primary Cervical Dystonia
Brief Title: Deep Brain Stimulation to Treat Cervical Dystonia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050222; 05-N-0222
Record Dates: First submitted 2005-08-18; First posted 2005-08-19 (Estimated); Last update posted 2006-07-06 (Estimated); Status verified 2006-07

CONDITIONS: Cervical Dystonia
Keywords: Spasmodic Torticollis; Treatment; Physiology; Surgery; Cervical Dystonia
MeSH Terms: conditions — Torticollis | interventions — Electrodes

INTERVENTIONS:
Device: Electrodes

SUMMARY:
This study will evaluate the effectiveness of deep brain stimulation (DBS) for treating primary dystonia. Patients with dystonia have muscle spasms that cause uncontrolled twisting and repetitive movement or abnormal postures. Medical therapies are available, but not all patients get adequate relief from the abnormal movements or the pain associated with them. DBS is a surgical procedure that interrupts neuronal circuits in the globus pallidus interna (Gpi) and subthalamic nucleus (STN) - areas of the basal ganglia of the brain that do not work correctly in patients with dystonia. This results in decreased movement and therefore may lessen patients' symptoms and pain. The study will also examine the physiology of dystonia and determine whether the treatment effects of DBS in the Gpi differ significantly from DBS of the STN.

Patients 18 years of age and older with primary cervical dystonia that does not respond to medical treatment or botulinum toxin (Botox) may be eligible for this study. Candidates are screened with blood and urine tests, chest x-ray, electrocardiogram, and magnetic resonance imaging (MRI, see below) of the brain.

Each participant undergoes the following tests and procedures:

* Magnetic resonance imaging. This procedure is done after implantation of the stimulators to verify position of the electrodes. MRI uses a magnetic field and radio waves to produce images of the brain. The patient lies on a table that is moved into the scanner (a narrow cylinder), wearing earplugs to muffle loud knocking and thumping sounds that occur during the scanning process. The procedure usually lasts about 45 to 90 minutes, during which the patient is asked to lie still for up to 15 minutes at a time.
* Transcranial magnetic stimulation. This procedure maps brain function. A wire coil is held on the scalp, and a brief electrical current is passed through the coil, creating a magnetic pulse that stimulates the brain. During the stimulation, the patient may be asked to tense certain muscles slightly or perform other simple actions. The stimulation may cause a twitch in muscles of the face, arm, or leg, and the patient may hear a click and feel a pulling sensation on the skin under the coil. During the stimulation, electrical activity of muscles is recorded with a computer, using electrodes attached to the skin with tape.
* Neurologic evaluation. Before and after DBS, the patient's dystonia is measured with a standardized rating scale called the Toronto Western Spasmodic Torticollis Scale (TWSTRS).
* DBS treatment. Patients are randomly assigned to have electrodes implanted in either the Gpi or STN area of the basal ganglia. The electrodes are what stimulate the brain in DBS therapy. Before surgery, a frame is secured to the patient's head, and an MRI scan is done. DBS involves making two small incisions and two small holes in the skull, opening the lining around the brain, locating the Gpi or STN, securing the electrodes in place, and connecting them to the pulse generator that is placed under the skin below the collar bone. In addition, during the surgery, the patient is asked to move certain muscles. The muscle activity is recorded to gain a better understanding of the physiology of movement. After surgery, MRI scans are done to confirm placement of the electrodes.
* Stimulation and evaluation. After surgery, patients' movements are evaluated during and after stimulation. The changes in movement and function are videotaped and scored according to a rating scale. The optimal stimulation settings are determined and the stimulators are adjusted accordingly.

Neurologic evaluations with the TWSTRS scale are repeated at 1, 2, 3, 6 and 12 months after surgery, and the stimulators are adjusted as needed. Some of the evaluations are videotaped.

DETAILED DESCRIPTION:
Objective: For patients with cervical dystonia who have failed medical therapy, stereotactic deep brain stimulation (DBS) of the globus pallidus interna (Gpi) or subthalamic nucleus (STN) can provide significant symptom improvement, but it is not known which site provides maximum benefit or the physiologic mechanisms by which these improvements may occur. The study goals are to determine if DBS of Gpi or STN provides significant clinical improvement in patients with primary cervical dystonia, whether the anatomic DBS site (if either) provides optimal improvement, and to gain deeper insight into the underlying pathophysiology of this disorder.

Study population: Adult patients with medically refractory primary cervical dystonia will make-up the study population. Patients with primary cervical dystonia suffer a wide range of symptoms including physical deformity, speech difficulties, swallowing dysfunction, visual problems, and intractable pain, which can result in an inability to care for themselves.

Design: We propose placing DBS electrodes (using microelectrode guidance) bilaterally into either the Gpi or STN of medically refractory cervical dystonia patients. Physiological studies will be performed and compared with clinical changes to understand the mechanism of action of DBS and underlying pathophysiology of cervical dystonia.

Outcome measures: Clinical effectiveness of DBS of the Gpi or STN will be measured by the Toronto Western Spasmodic Torticollis Scale and monitored over time to determine the effectiveness of DBS and if there is an ideal anatomic stimulation site. Electrophysiologic outcome measures will be obtained to determine the underlying pathophysiology of cervical dystonia, and the mechanism of action of DBS.

ELIGIBILITY:
* INCLUSION CRITERIA

To be eligible for entry into the study, candidates must meet all the following criteria:

* Patients 18 years of age or older with primary cervical dystonia.
* Patients who are refractory to medication (to medications including; levodopa, anticholinergics, benzodiazepines, Baclofen) and who are considered surgical candidates. Patients will be determined to have medical refractory dystonia after having been treated by at least two medications of two different groups at the maximum recommended dose for a duration of at least two months.
* In case of treatment by intrathecal Baclofen delivered by a pump, a change to oral Baclofen must be performed, so that the pump can be taken out.
* Patients must have primary (idiopathic) cervical dystonia.
* Patients must have a minimum TWSTRS of 20 on optimal medical therapy.
* Patients must be mentally competent to consent for entrance into the protocol at the time of admission, or have legal guardian consent for them.
* Patients must have a signed DPA for research purposes.

EXCLUSION CRITERIA

Candidates will be excluded if:

* The patient has had previous lesioning surgery including radiofrequency lesioning of deep nuclei (thalamus, pallidum, STN).
* The patient currently has a functioning and effective stimulator in deep brain nuclei (thalamus, pallidum, STN).
* The patient is not able to tolerate surgery, as determined by the preoperative evaluation.
* The patient has a coagulopathy demonstrated by an abnormal prothrombin time, activated partial thromboplastin time, or thrombocytopenia (platelet count less than 150,000 platelets/mm(3)).
* The patient has a contraindication to MR-imaging such as previous surgery that involved placement of metal objects that could cause tissue damage or produce image artifacts.
* The patient has another chronic neurologic disorder
* The patient is pregnant at the time of surgery.
* The patient has epilepsy.
* The patient does not have access to proper follow-up care at home may not be eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-08; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Jankovic J, Leder S, Warner D, Schwartz K. Cervical dystonia: clinical findings and associated movement disorders. Neurology. 1991 Jul;41(7):1088-91. doi: 10.1212/wnl.41.7.1088. PMID 2067638